CLINICAL TRIAL: NCT03526939
Title: DRIVE (DRug Use and Infections in ViEtnam) Project : Ending the HIV Epidemic Among Persons Who Inject Drugs in Hai Phong, Viet Nam
Brief Title: DRug Use and Infections in Hai Phong ViEtnam Among Persons Who Inject Drugs
Acronym: DRIVE
Status: Completed | Type: Observational
Sponsor: New York University (Other)
Collaborators: Hai Phong Medical University (Other); Université Montpellier (Other); Centre for Supporting Community Development Initiatives (SCDI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: GCO 15-1533
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: HIV; Hepatitis C; Mental Health
Keywords: Persons who inject drugs; HIV; Hepatitis C; Vietnam; Behavioral Intervention
MeSH Terms: conditions — Hepatitis C; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and plasma aliquots and dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV negative from RDS round 1: HIV negative PWID subjects from RDS round 1
- HIV negative from RDS round 2: HIV negative PWID subjects from RDS round 2
- HIV negative from RDS round 3: HIV negative PWID subjects from RDS round 3

SUMMARY:
The overarching purpose of the proposed research is to demonstrate that high coverage implementation of combined prevention and care using an innovative approach will end the HIV epidemic among PWID in Haiphong, Viet Nam.

DETAILED DESCRIPTION:
Injection drug use is driving HIV epidemics in low/middle-income countries in Eastern Europe, Central Asia and Southeast Asia. "Combined prevention and care", including needle/syringe programs (NSP), medication-assisted treatment for opiate dependence, and antiretroviral treatment, has greatly reduced HIV incidence among persons who inject drugs (PWID) in many high-income areas, to where the "HIV epidemics" among PWID have "ended." There is now the need for a convincing demonstration that an HIV epidemic can be ended in a low/middle income setting. The overarching purpose of the proposed research is to demonstrate that high coverage implementation of combined prevention and care using an innovative approach will end the HIV epidemic among PWID in Haiphong, Viet Nam. The researchers define "ending the epidemic" as reducing HIV incidence to 0.5/100 person-years at risk.

Data collection will include recruitment using repeated community based respondent driven sampling (RDS) surveys, once per year among PWID in Hai Phong. Participants will be given a quantitative questionnaire and tested for HIV and Hepatitis C (HCV). Peer support groups will be mobilized to help recruit PWID and assist in educations on the benefits of early ART, access to methadone, antiretroviral treatment and psychiatric services, and ways to prevent HIV and HCV transmission through safe injection practices and safe sex. Additionally, the investigators will develop large cohorts of HIV positive and HIV negative PWID to closely document behaviors trends, HIV incidence, and the obstacles of the access and retention in HIV care and methadone. It has been shown that it is possible to end HIV epidemics among PWID in several high income countries. This study will build upon the knowledge and results gained in high income settings to achieve viral suppression among HIV positive PWID and reduce HIV/HCV incidence in order to "end the HIV epidemic" among persons who inject drugs in Haiphong.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* capable of giving informed consent and participating in study activities
* history of drug injection (confirmed by visual inspection or subject knowledge of injecting procedures)
* currently using an injectable drug (heroin or methamphetamine
* confirmed by urine test), not on MMT at initial recruitment
* willingness to participate in follow up studies, and expecting to remain in Haiphong for 2 years

Exclusion Criteria:

* less than 18 years of age
* on MMT at initial recruitment
* refusal to participate in follow-up studies
* no history of drug injection
* not currently using injectable drug (heroin or methamphetamine)
* not capable of giving informed consent
* those not expecting to remain in Haiphong for at least 2 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Residents of Haiphong Vietnam who currently are injecting drugs (heroin or methamphetamine) and at least 18 years of age
Sampling Method: Probability Sample
Enrollment: 5546 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of HIV in the PWID population | up to 48 months
  Incidence of HIV in the PWID population to be calculated in person-years

SECONDARY OUTCOMES:
Number of participants with unsuppressed viral load | up to 48 months
  The number of HIV+ PWID with unsuppressed viral load in the strategic subpopulation
Cost-Effectiveness ratio as compared to baseline | baseline, 3 years, 7 years, 10 years, and 20 years
  C1 and C0 denote the total (discounted) costs of HIV prevention and treatment for PWID. H1 and H0 denote the total number of incident HIV infections. If T denotes the average lifetime cost of treating someone with HIV and D denotes the average number of disability-adjusted life years (DALYs) lost due to HIV infection, then the cost per DALY saved by the proposed interventions is the "cost-effectiveness ratio," R = (∆C - ∆H*T)/(∆H*D).
Incremental costs averted | up to 20 years
  Estimated incremental costs per HIV infection averted
Lifetime medical costs | up to 20 years
  Estimated lifetime medical costs for treating HIV infection

CONTACTS AND LOCATIONS:
Overall Officials: Don Des Jarlais, PhD, Principal Investigator — New York University
Locations (1):
- Haiphong Medical University, Haiphong, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Des Jarlais D, Khue PM, Feelemyer J, Arasteh K, Thi Huong D, Thi Hai Oanh K, Thi Giang H, Thi Tuyet Thanh N, Vinh VH, Heckathorn DD, Moles JP, Vallo R, Quillet C, Rapoud D, Michel L, Laureillard D, Hammett T, Nagot N. Using dual capture/recapture studies to estimate the population size of persons who inject drugs (PWID) in the city of Hai Phong, Vietnam. Drug Alcohol Depend. 2018 Apr 1;185:106-111. doi: 10.1016/j.drugalcdep.2017.11.033. Epub 2018 Feb 2. PMID 29432973
- [Background] Michel L, Des Jarlais DC, Duong Thi H, Khuat Thi Hai O, Pham Minh K, Peries M, Vallo R, Nham Thi Tuyet T, Hoang Thi G, Le Sao M, Feelemyer J, Vu Hai V, Moles JP, Laureillard D, Nagot N; DRIVE Study Team. Intravenous heroin use in Haiphong, Vietnam: Need for comprehensive care including methamphetamine use-related interventions. Drug Alcohol Depend. 2017 Oct 1;179:198-204. doi: 10.1016/j.drugalcdep.2017.07.004. Epub 2017 Aug 2. PMID 28800503
- [Background] Duong HT, Jarlais DD, Khuat OHT, Arasteh K, Feelemyer J, Khue PM, Giang HT, Laureillard D, Hai VV, Vallo R, Michel L, Moles JP, Nagot N; Drive Study Group. Risk Behaviors for HIV and HCV Infection Among People Who Inject Drugs in Hai Phong, Viet Nam, 2014. AIDS Behav. 2018 Jul;22(7):2161-2171. doi: 10.1007/s10461-017-1814-6. PMID 28612212
- [Background] Des Jarlais D, Duong HT, Pham Minh K, Khuat OH, Nham TT, Arasteh K, Feelemyer J, Heckathorn DD, Peries M, Moles JP, Laureillard D, Nagot N; (The Drive Study Team). Integrated respondent-driven sampling and peer support for persons who inject drugs in Haiphong, Vietnam: a case study with implications for interventions. AIDS Care. 2016 Oct;28(10):1312-5. doi: 10.1080/09540121.2016.1178698. Epub 2016 May 13. PMID 27178119
- [Background] Des Jarlais DC, Thi Huong D, Thi Hai Oanh K, Khue Pham M, Thi Giang H, Thi Tuyet Thanh N, Arasteh K, Feelemyer J, Hammett T, Peries M, Michel L, Vu Hai V, Roustide MJ, Moles JP, Laureillard D, Nagot N; DRIVE Study Team. Prospects for ending the HIV epidemic among persons who inject drugs in Haiphong, Vietnam. Int J Drug Policy. 2016 Jun;32:50-6. doi: 10.1016/j.drugpo.2016.02.021. Epub 2016 Feb 27. PMID 27006257
- [Background] Hammett TM, Trang NT, Oanh KTH, Huong NT, Giang LM, Huong DT, Nagot N, Des Jarlais DC. The relationship between health policy and public health interventions: a case study of the DRIVE project to "end" the HIV epidemic among people who inject drugs in Haiphong, Vietnam. J Public Health Policy. 2018 May;39(2):217-230. doi: 10.1057/s41271-017-0115-7. PMID 29531303